CLINICAL TRIAL: NCT02028013
Title: Management of Male Sexual Dysfunction With Bioresonance Technique, a New Egyptian Device
Brief Title: Management of Sexual Dysfunction With Bioresonance Technique
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Man Clinic for Andrology, Male Infertility and Sexual Dysfunction (Other)
Responsible Party: Principal Investigator, Khaled Abdulmoneim Gadalla, Dr, Man Clinic for Andrology, Male Infertility and Sexual Dysfunction
Other Study IDs: 002
Record Dates: First submitted 2014-01-03; First posted 2014-01-06 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Sexual Dysfunction; Erectile Dysfunction; Premature Ejaculation
Keywords: Erectile dysfunction, sexual dysfunction, bioresonance
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Erectile Dysfunction; Premature Ejaculation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Bioresonance is the big promise of the medical technology of the future because it stimulates the self-regenerating system of the body by affecting the body's most essential procedures. The big advantage is that its multiple and there are no harmful side effects. This therapy teaches something to the body what in a younger and healthier state it had already Bioresonance is based on the scientific principle that metabolism within cells is influenced by one's electromagnetic field.

We start to use bioresonance technology in management of erectile dysfunction , premature ejaculation, decreased libido.

ELIGIBILITY:
Inclusion Criteria:

* erectile dysfunction Premature ejaculation Decreased libido

Exclusion Criteria:

* nil

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients complaining from erectile dysfunction
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-07 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | 2-6 months

SECONDARY OUTCOMES:
Penile duplex study | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Khaled A Gadalla, MD, Principal Investigator — AlAzhar university , Man clinic
Locations (1):
- Man Clinic, Cairo, Egypt